CLINICAL TRIAL: NCT06302530
Title: "Effectiveness of the Ultrasound - Guided Lengthening of the Gastrocsoleus Complex"
Acronym: EUGLGC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCV/2022-2023/155
Record Dates: First submitted 2024-02-12; First posted 2024-03-08 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-04

CONDITIONS: Gastrocnemius Equinus
Keywords: Gastrocnemius lengthening; Equinus; Contracture correction surgery; ankle range of motion improvement; Orthopedic foot surgery

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: To reduce bias, the study will use double-blind blinding. Patients will not know the group to which they have been assigned. In addition, the assessors performing the ankle range of motion measurements by goniometry will be blinded to each patient's treatment group.
  Randomization to each group will be performed using opaque sealed envelopes that will be opened in the operating room just prior to surgery. Neither the surgeon nor the patient will know the assignment until that time.
  The statistical analysis will also be performed in a blinded manner, without the statistician knowing the intervention received by each group. Only after the analysis will the groups be unblinded.
  In this way, the aim is to reduce the possibility of knowledge of the assigned treatment influencing the evaluation of the results, both on the part of the patients and of the evaluators and analysts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group Strayer: (Experimental): This group will consist of patients with isolated gastrocnemius contracture who will be operated with the Strayer technique. This consists of ultrasound-guided surgical recession of the gastrocnemius tendon distally.
  Interventions: Procedure: Stayer
- Group Plantar transection: (Experimental): This group will include patients with mild contracture of the triceps suralis who will undergo surgery by ultrasound-guided transection of the plantar tendon on the medial aspect of the gastrocnemius.
  Interventions: Procedure: Plantar transection
- Group Bahuman (Experimental): This group will include patients undergoing an ultrasound-guided recession of the anterior gastrocnemius aponeurosis, where the myotendinous junction is accessed 3 cm proximally using saline for hydrodissection, followed by portal enlargement and scalpel introduction to transect the aponeurosis and plantar tendon under ultrasound verification, without requiring sutures, with patients wearing a Walker boot for 4 weeks and adhering to a stretching protocol
  Interventions: Procedure: Baumann
- Group Gastro-Soleus (Experimental): This group will include patients undergoing a modified Strayer technique involving the soleus. Under local anesthesia and ultrasound guidance, the gastrocnemius aponeurosis and a superficial portion of the soleus tendon will be transected
  Interventions: Procedure: Gastro-Soleus

INTERVENTIONS:
Procedure: Stayer — In group A, the intervention involves using the Strayer technique, an echo-guided recession of the gastrocnemius tendon, with local anesthesia and sedation as needed. The patient can be in a prone or supine position. Ultrasound will identify the sural nerve and blood vessels to prevent damage. The entry point is 2-3 cm distal to the medial head of the gastrocnemius. Local anesthetic is infiltrated, and blunt dissection creates a working space. V-shaped curettes widen the entry point without harming noble structures.
  Under direct ultrasound control, a curved scalpel is inserted until reaching the medial border of the gastrocnemius tendon. Transection occurs progressively from medial to lateral while flexing the foot. Verification of complete tendon transection is done with a blunt dissector. Finally, a dressing with adhesive strips and an elastic bandage is applied, eliminating the need for sutures.
  Arms: Group Strayer:
Procedure: Plantar transection — In group B, an echo-guided transection of the plantar tendon will be performed. Local anesthesia and sedation will be used as needed. The patient will be in prone or supine position. The plantar tendon will be identified ultrasonographically on the medial aspect of the gastrocnemius distal to the myotendinous junction. Local anesthetic will be infiltrated at that point to isolate the plantar tendon. An ultrasound-guided retrograde hook is introduced until the plantar tendon is engaged. Then proceed to retrograde transection of the tendon from lateral to medial, verifying complete section. At the end, a dressing with adhesive strips and elastic bandage, without sutures, will be performed.
  Arms: Group Plantar transection:
Procedure: Baumann — It consists of an ultrasound-guided recession of the anterior gastrocnemius aponeurosis. Under local anesthesia, the myotendinous junction is accessed 3 cm proximal to the myotendinous junction, using saline for hydrodissection. Under ultrasound guidance, the entry portal is enlarged and a scalpel is introduced for transection of the aponeurosis and plantar tendon. The procedure is verified with a buttoned probe and does not require sutures. The patient wears a Walker boot for 4 weeks and follows a stretching protocol.
  Arms: Group Bahuman
Procedure: Gastro-Soleus — This technique adapts the Strayer technique to include the soleus. Under local anesthesia, access is gained 4-5 cm distal to the medial head of the gastrocnemius. Transection of the gastrocnemius aponeurosis and a superficial section of the soleus tendon are performed, all under ultrasound guidance. Without the need for sutures, the patient wears a Walker boot for 4 weeks and follows a progressive rehabilitation protocol.
  Arms: Group Gastro-Soleus

SUMMARY:
The study analyzes the effectiveness of different ultrasound-guided surgical techniques to treat gastrocnemius contracture and equinus deformity, conditions that affect ankle dorsiflexion and can cause problems such as plantar fasciitis and metatarsalgia. Four techniques were compared: Strayer, Plantaris, Baumann and Gastro-soleo, evaluating their impact on the improvement of ankle motion.

DETAILED DESCRIPTION:
Equinus deformity is a common deformity caused by contracture of the triceps suralis, especially the gastrocnemius. This causes limitation of ankle dorsiflexion, pain and gait incompetence. Treatment includes surgical lengthening techniques such as gastrocnemius tendon recession (Strayer) or isolated plantar tendon transection.

The minimally invasive Strayer technique is effective but carries morbidity. Ultrasound-guided plantar tendon transection is a new minimally invasive technique but its effectiveness has not been well established.

The study will evaluate the effectiveness of four ultrasound-guided surgical techniques in improving ankle dorsiflexion in patients with equinus due to gastrocnemius contracture. The Strayer, Plantaris, Baumann, and Gastro-soleo techniques will be compared, analyzing their impact on mobility before and after surgery.

Patients will be assigned to different groups based on the applied technique, following specific inclusion and exclusion criteria for each procedure. For statistical analysis, Wilcoxon and paired Student's t-tests will be used, depending on data distribution. Additionally, a repeated-measures ANOVA with Tukey's post-hoc tests will be applied to compare the results between techniques and determine which achieves the greatest increase in dorsiflexion range.

All techniques are expected to significantly improve dorsiflexion, with differences in the magnitude of change. The Gastro-soleo technique is anticipated to show the highest absolute increase, while Strayer may be the most statistically effective.

The study complies with ethical requirements and has the approval of the ethics committee of the Catholic University of Valencia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological diagnosis of clubfoot.
* Limitation of passive dorsiflexion of the ankle (<10°).
* Associated pain and functional limitation
* Absence of previous ankle/foot surgeries

Exclusion criteria:

* Neurologic or congenital disease.
* Advanced ankle joint osteoarthritis
* Peripheral vascular insufficiency
* Uncontrolled diabetes mellitus
* Severe hepatic or renal disease
* Coagulopathies or anticoagulant therapy

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Ankle range of motion | Pre-surgery, 2 months, 6months and 1 year.
  Measurement in degrees of the passive dorsiflexion range of the ankle using a goniometer, with the patient in supine position and knee extended.

SECONDARY OUTCOMES:
Visual Analog Scale. | Pre-surgery,2 months,6months and 1 year.
  This is a measurement tool used to evaluate the intensity of symptoms such as pain, where the patient marks on a visual line the perceived intensity, being 0 no pain and 10 a lot of pain.
American Orthopedic Foot and Ankle Score | Pre-surgery,2 months,6months and 1 year.
  The AOFAS Ankle-Hindfoot Scale was designed by the American Foot and Ankle Society to provide an international method to assess the clinical status of the ankle and foot.
  This questionnaire incorporates subjective and objective factors that are scored using a numerical scale and describe variables of function, alignment and pain. The score ranges from 0 to 100 depending on the degree of limitation of the patient.
Complications | Pre-surgery,2 months,6months and 1 year.
  Record of complications related to surgery.

CONTACTS AND LOCATIONS:
Overall Officials: SIMONE MORONI, Dr., Principal Investigator — UNIVERSIDAD CATOLICA DE VALENCIA; JAVIER FERRER-TORREGROSA, Dr., Study Director — UNIVERSIDAD CATOLICA DE VALENCIA
Locations (3):
- Spain (3):
  - Podologia Avançada, Granollers, Barcelona
  - Clinica Mayral foot center, Barcelona, Barcelon
  - Clinica Pasito a pasito, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cychosz CC, Phisitkul P, Belatti DA, Glazebrook MA, DiGiovanni CW. Gastrocnemius recession for foot and ankle conditions in adults: Evidence-based recommendations. Foot Ankle Surg. 2015 Jun;21(2):77-85. doi: 10.1016/j.fas.2015.02.001. Epub 2015 Feb 26. PMID 25937405
- [Background] DiGiovanni CW, Kuo R, Tejwani N, Price R, Hansen ST Jr, Cziernecki J, Sangeorzan BJ. Isolated gastrocnemius tightness. J Bone Joint Surg Am. 2002 Jun;84(6):962-70. doi: 10.2106/00004623-200206000-00010. PMID 12063330
- [Background] Barouk P, Barouk LS. Clinical diagnosis of gastrocnemius tightness. Foot Ankle Clin. 2014 Dec;19(4):659-67. doi: 10.1016/j.fcl.2014.08.004. Epub 2014 Sep 26. PMID 25456715
- [Background] Maluf KS, Mueller MJ, Strube MJ, Engsberg JR, Johnson JE. Tendon Achilles lengthening for the treatment of neuropathic ulcers causes a temporary reduction in forefoot pressure associated with changes in plantar flexor power rather than ankle motion during gait. J Biomech. 2004 Jun;37(6):897-906. doi: 10.1016/j.jbiomech.2003.10.009. PMID 15111077
- [Background] STRAYER LM Jr. Recession of the gastrocnemius; an operation to relieve spastic contracture of the calf muscles. J Bone Joint Surg Am. 1950 Jul;32-A(3):671-6. No abstract available. PMID 15428491
- [Background] Kindred KB, Kapsalis AP, Adams WJE, Miller JM, Blacklidge DK, Elliott BG, Hoffman SM. The Role of the Plantaris in Intramuscular Gastrocnemius Equinus Correction. J Foot Ankle Surg. 2023 Mar-Apr;62(2):272-274. doi: 10.1053/j.jfas.2022.07.006. Epub 2022 Jul 30. PMID 36096902
- [Background] Hickey B, Lee J, Stephen J, Antflick J, Calder J. It is possible to release the plantaris tendon under ultrasound guidance: a technical description of ultrasound guided plantaris tendon release (UPTR) in the treatment of non-insertional Achilles tendinopathy. Knee Surg Sports Traumatol Arthrosc. 2019 Sep;27(9):2858-2862. doi: 10.1007/s00167-019-05451-0. Epub 2019 Mar 7. PMID 30847522
- [Background] Moroni S, Fernandez-Gibello A, Nieves GC, Montes R, Zwierzina M, Vazquez T, Garcia-Escudero M, Duparc F, Moriggl B, Konschake M. Anatomical basis of a safe mini-invasive technique for lengthening of the anterior gastrocnemius aponeurosis. Surg Radiol Anat. 2021 Jan;43(1):53-61. doi: 10.1007/s00276-020-02536-1. Epub 2020 Jul 23. PMID 32705404